CLINICAL TRIAL: NCT06806592
Title: A Double Blind, Randomised, Placebo-controlled Trial Evaluating the Efficacy and Safety of Nerandomilast Over at Least 26 Weeks in Patients With Systemic Autoimmune Rheumatic Diseases Associated Interstitial Lung Diseases (SARD-ILD)
Brief Title: A Study to Test Whether Nerandomilast Helps People With Lungfibrosis Related to Rheumatic Diseases
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1305-0046; 2024-512849-17-00 (Registry Identifier: CTIS); U1111-1305-5857 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2025-01-28; First posted 2025-02-04 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Interstitial Lung Diseases; Systemic Autoimmune Rheumatic Diseases Associated Interstitial Lung Diseases
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nerandomilast (Experimental): Participants with SARD-ILDs will receive nerandomilast.
  Interventions: Drug: Nerandomilast
- Placebo (Placebo Comparator): Participants with SARD-ILDs will receive placebo.
  Interventions: Drug: Placebo matching nerandomilast

INTERVENTIONS:
Drug: Nerandomilast — Nerandomilast
  Other Names: JASCAYD®
  Arms: Nerandomilast
Drug: Placebo matching nerandomilast — Placebo matching nerandomilast
  Arms: Placebo

SUMMARY:
Adults 18 years of age and older or above legal age with lung fibrosis related to systemic autoimmune rheumatic disease can participate in this study. People can only take part if they show no improvement in lung function after standard treatment with immunosuppressant medicine. The main purpose of this study is to find out how a medicine called nerandomilast affects the lungs in people with systemic autoimmune rheumatic disease.

Participants are put into 2 groups randomly, which means by chance. One group takes nerandomilast tablets and the other group takes placebo tablets. Placebo tablets look like nerandomilast tablets but do not contain any medicine. Participants take a tablet 2 times a day for at least 26 weeks and up to 1 year. Participants continue immunosuppressant treatment for their underlying rheumatic disease.

Participants are in the study for about 7.5 to 13 months depending on when they join the study. During this time, they visit the study site about 9 to 10 times. At study visits, participants have lung function tests. At select visits, chest imaging is performed. Participants fill in questionnaires about their symptoms and quality of life. The results between the 2 groups are compared to see whether the treatment works. The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria :

* Participant has systemic autoimmune rheumatic diseases associated interstitial lung diseases (SARD-ILD), defined as

  * Diagnosis by a rheumatologist with at least 1 of the following SARDs: Rheumatoid arthritis (RA), systemic sclerosis (SSc) (participants must be anticentromere auto-antibody negative), idiopathic inflammatory myopathy (IIM), Sjögren's disease, or Mixed connective tissue disease (MCTD)
  * Presence of fibrotic interstitial lung disease (ILD) on high-resolution computed tomography (HRCT), defined as presence of reticular abnormality with traction bronchiectasis with or without honeycombing (HC), with disease extent >10% on HRCT performed within 12 months of Visit 1 or, if historical scan is not available, on baseline HRCT taken prior to Visit 2, as confirmed by central review
* No lung function improvement and no clinically significant ILD improvement as a treatment response to immunosuppressant (IS) therapy according to both criteria:

  * No improvement in absolute forced vital capacity (FVC) % predicted >5% within the 15 months prior to Visit 1, as measured by 2 spirometry assessments that must be ≥3 months apart. (Note: Visit 1 spirometry may be used to fulfill the inclusion criterion if there is only 1 spirometry reading in the 15 months prior to Visit 1)
  * No clinically significant improvement in ILD based on clinician's judgement (including symptoms, imaging/HRCT, or other assessments as considered relevant and documented by the Investigator)
* FVC ≥45% of predicted normal at Visit 1
* Diffusing capacity of the lungs for carbon monoxide (DLCO) ≥25% of predicted normal corrected for haemoglobin (Hb) within 3 months prior to or at Visit 1
* Participants must be on stable treatment with any IS agent for ≥6 months (or ≥3 months for participants with IIM-ILD) with the following specifications:

  * If using prednisone, participants must be on stable dose for ≥4 weeks prior to Visit 2
  * If using rituximab, participants must have completed their first cycle >6 months prior to Visit 2
* If using nintedanib, participants must be on a stable dose for ≥12 weeks prior to Visit 2
* In the opinion of the Investigator, no change in background standard of care (SoC) treatment with immunosuppressant (IS), immunomodulator (IM), or nintedanib is planned
* Further inclusion criteria apply

Exclusion Criteria :

* Organising pneumonia as predominant pattern in the HRCT
* Prebronchodilator forced expiratory volume in 1 second (FEV1)/ forced vital capacity (FVC) <0.7 at Visit 1
* Acute ILD exacerbation within 3 months prior to Visit 1 and/or during the screening period, based on Investigator judgement
* Active vasculitis, unstable or uncontrolled within 8 weeks prior to Visit 1 or during the screening period
* Any suicidal behaviour in the past 2 years
* Any suicidal ideation of type 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) in the past 3 months or at Visit 1, and/or at Visit 2
* Use of any of the following medications: cyclophosphamide within 6 months of Visit 1, pirfenidone within 8 weeks of Visit 1
* Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-09-13 (Actual); Primary Completion 2027-07-17 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Absolute change from baseline in quantitative interstitial lung disease (QILD) score [%] on high-resolution computed tomography (HRCT) at Week 26 | At baseline and at Week 26
  QILD will be assessed via quantitative high-resolution computed tomography (qHRCT). QILD are quantitative measures of different radiological patterns associated with lung fibrosis. QLF is a measure of reticulation with architectural distortion. QGGO is a measure of ground glass opacities (i.e. hazy or cloudy areas) within the lung. QHC is a measure of HC within the lung. QILD is the sum of QLF, QGGO, and QHC.
  Quantification of HRCT scans will be performed centrally via a machine learning algorithm. QILD [%] is the QILD volume [mL] as a percent of the total lung volume.
  A higher QILD percentage or volume indicates a higher extent of disease.

SECONDARY OUTCOMES:
Absolute change from baseline in quantitative lung fibrosis (QLF) score [%] on HRCT at Week 26 | At baseline and at Week 26
  QLF will be assessed via qHRCT. QLF are quantitative measures of different radiological patterns associated with lung fibrosis. QLF is a measure of reticulation with architectural distortion.
  Quantification of HRCT scans will be performed centrally via a machine learning algorithm. QILD [%] is the QILD volume [mL] as a percent of the total lung volume.
  A higher QILD percentage or volume indicates a higher extent of disease.
Absolute change from baseline in quantitative ground glass opacity (QGGO) score [%] on HRCT at Week 26 | At baseline and at Week 26
  QGGO will be assessed via qHRCT. QGGO are quantitative measures of different radiological patterns associated with lung fibrosis. QGGO is a measure of ground glass opacities (i.e. hazy or cloudy areas) within the lung.
  Quantification of HRCT scans will be performed centrally via a machine learning algorithm.
  A higher QGGO percentage or volume indicates a higher extent of disease.
Absolute change from baseline in vascular volume [%] on HRCT at Week 26 | At baseline and at Week 26
Absolute change from baseline in forced vital capacity (FVC) [mL] at Week 26 | At baseline and at Week 26
  FVC will be assessed using standardised spirometry equipment which will be provided centrally with supplies of precalibrated disposable flow sensors. Spirometry will be conducted with the participant in a seated position. It is preferable that the same trained individual (i.e. PFT specialist or pulmonologist) performs the PFTs for a given participant. The best of 3 efforts will be defined as the highest FVC obtained on any of three blows meeting the 2019 American Thoracic Society/European Respiratory Society (ATS/ERS) criteria (with a maximum of eight attempts). Predicted normal values will be calculated according to global lung function initiative (GLI).
Absolute change from baseline in supplemental oxygen use over the whole trial for oxygen users at baseline | At baseline and at Week 52
Time to first supplemental oxygen use during the trial for oxygen non-users at baseline | Up to Week 52
Occurrence of infection-related adverse events (AEs) from baseline over the duration of the trial | Up to 1 year

CONTACTS AND LOCATIONS:
Locations (157):
- United States (33):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic-Arizona, Scottsdale, Arizona
  - University of California Los Angeles, Los Angeles, California
  - Paradigm Clinical Research - San Diego, San Diego, California
  - National Jewish Health, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Meris Clinical Research-Brandon-69466, Brandon, Florida
  - Miami VA Healthcare System, Miami, Florida
  - Piedmont Physicians Pulmonary & Sleep Medicine of Buckhead, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Northshore University Health System, Evanston, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - LSU Health Sciences Center, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Northwell Health, Great Neck, New York
  - NYU Langone Health, New York, New York
  - Columbia University Medical Center-New York Presbyterian Hospital, New York, New York
  - Onsite Clinical Solutions, Salisbury, North Carolina
  - Southeastern Research Center-Winston Salem-69289, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Temple Lung Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - Rheumatology and Pulmonary Clinic, Beckley, West Virginia
  - University of Wisconsin, Madison, Wisconsin
- Australia (5):
  - Royal Prince Alfred Hospital, Camperdown, Sydney, New South Wales
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - Austin Hospital, Heidelberg, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Austria (3):
  - Krems University Hospital, Krems
  - AKH - Medical University of Vienna, Vienna
  - Klinikum Wels - Grieskirchen GmbH, Wels
- China (17):
  - Beijing Chao-Yang Hospital, Beijing
  - China-Japan Friendship Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - West China Hospital, Sichuan University, Chengdu
  - People's Hospital of Sichuan Province, Chengdu
  - Guangdong Provincial People's Hospital, Guangzhou
  - The First Affiliated Hospital, Zhejiang University, Hangzhou
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang
  - University Hospital_Macau University of Science and Technology, Macau
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Huashan Hospital, Fudan University, Shanghai
  - Tianjin Medical University General Hospital, Tianjin
  - Wuhan Union Hospital, Wuhan
  - Tongji Hospital Affiliated Tongji Medical College Huazhong University of S & T, Wuhan
  - First Affiliated Hospital of Xiamen University, Xiamen
  - Zhuzhou Central Hospital, Zhuzhou
- France (8):
  - HOP d'Angers, Angers
  - HOP Pellegrin, Bordeaux
  - Hôpital Claude Huriez, Lille
  - Hôpital Cochin, Paris
  - HOP Bichat, Paris
  - HOP Sud, Rennes
  - HOP Civil, Strasbourg
  - Hôpital Rangueil - CHU de Toulouse, Toulouse
- Germany (19):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Immanuel-Krankenhaus GmbH, Berlin
  - Universitätsklinikum Bonn AöR, Bonn
  - Städtisches Klinikum Braunschweig gGmbH, Braunschweig
  - Gesundheit Nord gGmbH | Klinikverbund Bremen, Bremen
  - Krankenhaus Porz am Rhein gGmbH, Cologne
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Erlangen, Erlangen
  - Ruhrlandklinik, Westdeutsches Lungenzentrum am Universitätsklinikum Essen gGmbH, Essen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Helios Fachklinik Vogelsang-Gommern GmbH, Gommern
  - Medizinische Hochschule Hannover, Hanover
  - St. Elisabeth Gruppe GmbH Katholische Kliniken Rhein-Ruhr, Herne
  - medius Kliniken gGmbH, Kirchheim unter Teck
  - Klinikum Konstanz, Konstanz
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck
  - Johannes Wesling Klinikum Minden, Minden
  - Klinikum der Universität München AÖR, München
  - Krankenhaus Barmherzige Brüder Regensburg, Regensburg
- Italy (8):
  - ASST degli Spedali Civili di Brescia, Brescia
  - A. O. Universitaria Careggi, Florence
  - Fondazione IRCCS Ca'Granda-Ospedale Maggiore Policlinico, Milan
  - Ospedale San Raffaele S.r.l., Milan
  - Azienda Ospedaliero-Universitaria di Modena, Modena
  - Azienda Ospedaliera Universitaria di Padova, Padua
  - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - AOU Policlinico Umberto I, Roma
- Japan (15):
  - Fujita Health University Hospital, Aichi, Toyoake
  - Hospital of the University of Occupational and Environmental Health, Fukuoka, Kitakyushu
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - Sapporo Medical University Hospital, Hokkaido, Sapporo
  - Hokkaido University Hospital, Hokkaido, Sapporo
  - Kagawa University Hospital, Kagawa, Kita-gun
  - St. Marianna University Hospital, Kanagawa, Kawasaki
  - Kitasato University Hospital, Kanagawa, Sagamihara
  - Kyoto University Hospital, Kyoto, Kyoto
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Osaka Medical and Pharmaceutical University Hospital, Osaka, Takatsuki
  - Saitama Medical University Hospital, Saitama, Iruma-gun
  - Juntendo University Hospital, Tokyo, Bunkyo-Ku
  - Nippon Medical School Hospital, Tokyo, Bunkyo-ku
  - Keio University Hospital, Tokyo, Shinjuku-ku
- Mexico (7):
  - Investigacion y Biomedicina de Chihuahua S.C., Chihuahua City
  - Centro Integral en Reumatologia, SA. de CV., Guadalajara
  - Soltmed Smo, Mexico City
  - CITER Centro de Investigación y Tratamiento de las Enfermedades Reumaticas SA de CV, Mexico City
  - Inst Nac de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City
  - Medical Care & Research SA de CV, Mérida
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Monterrey
- Netherlands (3):
  - Zuyderland Medisch Centrum, Heerlen
  - St. Antonius Ziekenhuis, Nieuwegein
  - Erasmus Medisch Centrum-ROTTERDAM-50697, Rotterdam
- Norway (2):
  - Akershus Universitetssykehus HF, Nordbyhagen
  - Sykehuset Telemark HF, Avd. Skien, Skien
- GCM Medical Group, PSC, San Juan, Puerto Rico
- South Korea (4):
  - Seoul National University Bundang Hospital, Seongnam
  - Kyung Hee University Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Soonchunhyang University Hospital Seoul, Seoul
- Spain (14):
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital de Basurto, Bilbao
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Juan Ramón Jimenez, Huelva
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clínico de Santiago, Santiago de Compostela
  - Hospital Universitario Virgen De La Macarena, Seville
  - Hospital Virgen del Rocío, Seville
  - Hospital Dr. Peset, Valencia
  - Complejo Hospitalario Universitario de Vigo, Vigo
- Switzerland (6):
  - Cantonal Hospital of Aarau, Aarau
  - Universitätsspital Basel, Basel
  - Hopitaux Universitaires de Geneve (HUG), Geneva
  - Neuchatel Hospital Network, Neuchâtel
  - Kantonsspital St.Gallen, Sankt Gallen
  - University Hospital Zurich, Zurich
- United Kingdom (12):
  - Antrim Area Hospital, Antrim
  - Royal United Hospital, Bath, Bath
  - Heartlands Hospital, Birmingham
  - Chapel Allerton Hospital, Leeds
  - St George's Hospital-London-26733, London
  - University College Hospital, London
  - Altnagelvin Area Hospital, Londonderry
  - Luton & Dunstable University Hospital, Luton
  - NIHR Lancashire Clinical Research Facility, Preston
  - Northern General Hospital, Sheffield
  - Royal Cornwall Hospital, Truro
  - Southend University Hospital, Westcliffe-on-Sea

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "time frame" are fulfilled, researchers can use the following link https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents -upon signing of a "Document Sharing Agreement". For study data -1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.clinicalstudies.boehringer-ingelheim.com/msw/datatransparency